CLINICAL TRIAL: NCT00002662
Title: PHASE III COMPARISON OF TAXOTERE (DOCETAXEL) AND TAXOL (PACLITAXEL) IN PATIENTS WITH ADVANCED BREAST CANCER
Brief Title: Paclitaxel or Docetaxel in Treating Women With Advanced Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aventis Pharmaceuticals (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: AVENTIS-56976-TAX-311; CDR0000064232 (Registry Identifier: PDQ (Physician Data Query)); RP-56976-TAX-311; NCI-V95-0680
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2004-04

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; stage IIIA breast cancer; recurrent breast cancer; stage IIIB breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Paclitaxel

INTERVENTIONS:
Drug: docetaxel
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known whether paclitaxel is more effective than docetaxel for breast cancer.

PURPOSE: Randomized phase III trial to study the effectiveness of paclitaxel or docetaxel in treating women with stage IIIB or metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the response rate in women with metastatic or locally advanced, inoperable adenocarcinoma of the breast treated with docetaxel vs paclitaxel.
* Compare the toxicity of these regimens in these patients.
* Compare the time to disease progression, duration of response, quality of life, and survival of patients treated with these regimens.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive docetaxel IV over 1 hour on day 1. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive paclitaxel IV over 3 hours on day 1. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline and after courses 4 and 6.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 400 patients (200 per arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven metastatic or locally advanced, inoperable adenocarcinoma of the breast

  * Clinically evident metastases (e.g., clearly malignant lesions on chest x-ray or CT or abdominal CT do not require histologic confirmation)
  * Hot spots on bone scan not shown to be malignant on plain x-rays are not adequate evidence of malignant disease in the absence of other lesions
* Must meet 1 of the following conditions:

  * Disease progression after 1 prior chemotherapy regimen for locally advanced or metastatic disease (which may or may not have followed a separate adjuvant regimen using chemotherapy or hormonal therapy)
  * Locally advanced or metastatic disease during or after 1 adjuvant or neoadjuvant chemotherapy regimen
  * One of the above chemotherapy regimens must have contained an anthracycline (e.g., doxorubicin, but not mitoxantrone)
  * Single drug substitution (e.g., methotrexate for doxorubicin) during prior combination chemotherapy allowed
* Bidimensionally measurable
* No clinical or radiographic evidence of brain or leptomeningeal disease
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Sex:

* Female

Menopausal status:

* Not specified

Performance status:

* Karnofsky 60-100% OR
* ECOG 0-2

Life expectancy:

* At least 12 weeks

Hematopoietic:

* Absolute neutrophil count at least 2,000/mm3
* Platelet count at least 100,000/mm3

Hepatic:

* Bilirubin normal
* SGOT no greater than 2.5 times upper limit of normal

Renal:

* Creatinine no greater than 2.0 mg/dL
* No uncontrolled hypercalcemia

Cardiovascular:

* No myocardial infarction within the past 6 months
* No history of arrhythmia requiring treatment
* No heart block
* No clinical evidence of congestive heart failure
* No unstable angina (e.g., new onset, crescendo, or rest angina)
* Stable exertional angina allowed

Other:

* No current symptomatic grade 2 or greater peripheral neuropathy
* No history of hypersensitivity to products containing Cremophor EL (e.g., cyclosporine or teniposide) or Polysorbate 80 (e.g., IV etoposide)
* No serious infection
* No significant psychiatric disease that would preclude study
* No other malignancy within the past 5 years except nonmelanomatous skin cancer or completely excised carcinoma in situ of the cervix
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior bone marrow or stem cell transplantation

Chemotherapy:

* See Disease Characteristics
* At least 3 weeks since prior chemotherapy (2 weeks for oral cyclophosphamide or 6 weeks for nitrosoureas or mitomycin)
* No prior high-dose chemotherapy given with ablative intent
* No prior taxoids
* No other concurrent antineoplastic therapy

Endocrine therapy:

* See Disease Characteristics
* Prior hormonal therapy as adjuvant therapy or for metastatic disease allowed
* At least 1 week since prior hormonal therapy
* No concurrent corticosteroids except:

  * Prophylaxis or treatment for acute hypersensitivity reactions
  * Chronic therapy (more than 6 months) at low doses (20 mg/day or less of methylprednisolone or equivalent)

Radiotherapy:

* At least 4 weeks since prior radiotherapy to major bone marrow areas
* No prior high-dose radiotherapy given with ablative intent
* No concurrent radiotherapy except limited palliative radiotherapy (e.g., for a solitary rib fracture) during objective response

Surgery:

* See Disease Characteristics
* More than 2 weeks since prior surgery except simple biopsy or placement of venous access device

Other:

* At least 4 weeks since prior investigational drugs
* Concurrent medications known to alter cardiac conduction (e.g., digoxin, beta blockers, or calcium channel blockers) allowed
* No concurrent ketoconazole
* No concurrent bisphosphonates unless initiated more than 3 months before randomization
* No concurrent experimental drug or therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1994-08; Study Completion 2004-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter M. Ravdin, MD, Study Chair — The University of Texas Health Science Center at San Antonio
Locations (32):
- United States (32):
  - Montclair Regional Cancer Center, Birmingham, Alabama
  - Highlands Oncology Group, P.A. - Fayetteville, Fayetteville, Arkansas
  - Northeast Arkansas Clinic, Jonesboro, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - California Cancer Care, Inc., Greenbrae, California
  - Green Cancer Center at Scripps Clinic, La Jolla, California
  - Sidney Kimmel Cancer Center, San Diego, California
  - University of Colorado Cancer Center at University of Colorado Health Sciences Center, Denver, Colorado
  - Norwich Cancer Center, Norwich, Connecticut
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - Baptist Regional Cancer Institute - Jacksonville, Jacksonville, Florida
  - Georgia Cancer Specialists - DeKalb, Decatur, Georgia
  - Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Maine Center for Cancer Medicine and Blood Disorders - Scarborough, Scarborough, Maine
  - Tufts - New England Medical Center, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Southfield Oncology Institute, Inc., Southfield, Michigan
  - Mercy Arch Hematology Oncology, P.C., St Louis, Missouri
  - Carolinas Hematology-Oncology Associates, Charlotte, North Carolina
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Hematology Oncology Consultants Inc, Columbus, Ohio
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Oncology-Hematology Associates, Philadelphia, Pennsylvania
  - Roger Williams Medical Center, Providence, Rhode Island
  - Greenville Hospital System, Greenville, South Carolina
  - Baptist Regional Cancer Center - Knoxville, Knoxville, Tennessee
  - Charles A. Sammons Cancer Center, Dallas, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin